CLINICAL TRIAL: NCT04155320
Title: Provider-Assisted HIV Partner Notification & Testing With Prisoners in Indonesia: A Randomized Controlled Trial
Brief Title: Impart: Provider-Assisted HIV Partner Notification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Indonesia University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Gabriel John Culbert, Assistant Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2018-0754; R34MH115779 (NIH)
Record Dates: First submitted 2019-11-05; First posted 2019-11-07 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: HIV Infections; Partner Communication
Keywords: contact tracing; HIV prevention; partner notification
MeSH Terms: conditions — HIV Infections | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor is blinded as to treatment allocation during analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Subjects are encouraged to disclose their HIV status to their partner(s) with or without a counselor present (Options 1 & 2).
  Interventions: Behavioral: Standard Care
- Group B (Experimental): Subjects may choose to notify their partners themselves, with or without a counselor present (Options 1 & 2), or choose to have one or more partners notified anonymously by project staff (Option 3).
  Interventions: Behavioral: IMPART

INTERVENTIONS:
Behavioral: IMPART — Subjects receive counseling about partner notification and are assisted in identifying all their partners and choosing a notification method for each partner. Subjects have the option to: 1) disclose their HIV status to their partner(s) by themselves (self-tell), 2) disclose their HIV status to their partner(s) with a healthcare provider present (tell together), or 3) have their partner(s) notified confidentially by a disease notifier (anonymous provider referral), who will locate partners, notify them of potential HIV exposure, and offer them HIV testing. Partners with an initial reactive HIV screening test will be referred to care and treatment services.
  Arms: Group B
Behavioral: Standard Care — Subjects receive counseling about partner notification and are assisted in identifying all their partners and choosing a notification method for each partner. Subjects are responsible for contacting and notifying their partner(s) on their own. Subjects have the option to: 1) disclose their HIV status to their partner(s) by themselves (self-tell) or 2) disclose their HIV status to their partner(s) with a healthcare provider present (tell together). Subjects may decide which partners to notify and may choose the same or a different method for each partner.
  Arms: Group A

SUMMARY:
Researchers will conduct a 2-arm pilot randomized controlled trial with HIV-infected index patients recruited from two all-male prisons in Indonesia to assess the acceptability and feasibility of provider-assisted HIV partner notification (provider referral) and examine its potential to increase the number of partners who are tested for HIV and subsequently linked to prevention and treatment services.

DETAILED DESCRIPTION:
This study compares three options for partner notification:

* Option 1 (Self-tell): Participant is encouraged to disclose his HIV+ status to his partner(s) and given information about sites where his partner(s) can receive free HIV testing.
* Option 2 (Tell together): Participant discloses his HIV+ status to his partners with a counselor (project staff) present. Counselor refers the partner to HIV testing, including a study-affiliated HIV testing site.
* Option 3 (Provider referral): Project staff (nurse or peer educator) will notify the partner anonymously - without identifying the participant (index patient). Partners are offered immediate HIV testing in their home or at a study-affiliated HIV testing site.

ELIGIBILITY:
Inclusion Criteria for HIV-positive Prisoners (N=65): Index patients must beat least 18 years of age, HIV-seropositive and aware of their HIV+ status; (HIV-infection documented by a rapid HIV test); sexually active and/or sharing needles in the 12 months before incarceration; incarcerated within the past 3 years and ≥6 months of their prison sentence remaining. We will limit enrollment to index patients who are willing to notify partners and have 1 or more partner(s) who have not yet been notified.

Inclusion Criteria for Partners: Eligible partners will be persons who participants (index patients) are able to identify by first and/or last name, residential address and/or mobile phone number, and physical descriptors (e.g., approximate height) and have given nurses permission to contact. No named partner will be excluded on the basis of religion, ethnicity, age, sex, or gender identity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2020-01-27 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-11-12 (Actual)

PRIMARY OUTCOMES:
Notified | 6 weeks from index patient enrollment
  Number of partners who are notified of shared HIV exposure
Tested | 6 weeks from index patient enrollment
  Number of partners who receive HIV testing subsequent to notification
Diagnosed | 6 weeks from index patient enrollment
  Number of partners who are HIV diagnosed subsequent to testing

SECONDARY OUTCOMES:
Linked to Care | 6 weeks from index patient enrollment
  Number of partners who have been evaluated for treatment by a physician subsequent to diagnosis
Initiated ART | 6 weeks from index patient enrollment
  Number of partners who have initiated antiretroviral therapy (ART) subsequent to linkage to care

CONTACTS AND LOCATIONS:
Locations (1):
- Rutan Cipinang, Jakarta Pusat, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Culbert GJ, Levy JA, Steffen AD, Waluyo A, Earnshaw VA, Rahadi A. Impart: findings from a prison-based model of HIV assisted partner notification in Indonesia. J Int AIDS Soc. 2023 Jun;26(6):e26132. doi: 10.1002/jia2.26132. PMID 37339342